CLINICAL TRIAL: NCT01767805
Title: Impact of Culture Conditions on the Embryo Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Thomas D'Hooghe, Prof. Dr., University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ML4563
Record Dates: First submitted 2013-01-08; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Embryo Development
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type of incubator (Other): Embryos are cultured in a standard incubator or a mini-incubator
  Interventions: Procedure: Standard incubator; Procedure: Mini incubator
- Oxygen concentration (Other): Embryos are cultured in an incubator with a gas mixture with 20% oxygen or with 5% oxygen
  Interventions: Procedure: 5% oxygen; Procedure: 20% oxygen

INTERVENTIONS:
Procedure: Standard incubator
  Arms: Type of incubator
Procedure: Mini incubator
  Arms: Type of incubator
Procedure: 5% oxygen
  Arms: Oxygen concentration
Procedure: 20% oxygen
  Arms: Oxygen concentration

SUMMARY:
The purpose of this study is to compare different culture conditions. The effect of the type of incubator (standard versus mini-incubator) and the effect of the oxygen concentration (5% versus 20%) will be evaluated on the embryo quality

ELIGIBILITY:
Inclusion Criteria:

* embryos of patients younger than 36 years old

Exclusion Criteria:

* embryos of patients older than 36 years old

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 790 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
embryo quality | day 1- day 3

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University Hospital Leuven, Catholic University Leuven, Leuven, Leuven
  - University Hospital Leuven, Catholic University Leuven, Leuven